CLINICAL TRIAL: NCT06755814
Title: Community-acquired Pneumonia in Immunosuppressed Adult Patients: Observational, Perspective Study, ItAlian ReGistry Of pNeumoniA in immUnocompromised paTients (ARGONAUT)
Brief Title: ItAlian ReGistry Of pNeumoniA in immUnocompromised paTients (ARGONAUT)
Acronym: ARGONAUT
Status: Recruiting | Type: Observational
Sponsor: Societa Italiana di Pneumologia (Other)
Responsible Party: Sponsor
Other Study IDs: 4656/ 2024
Record Dates: First submitted 2024-11-19; First posted 2025-01-01 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2024-12

CONDITIONS: Community Acquired Pneumonia (CAP)
Keywords: CAP; Immunosuppressed; Immunocompromised; Pneumonia; community-acquired pneumonia;
MeSH Terms: conditions — Community-Acquired Pneumonia; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood Serum Sputum BAL (bronchoalveolar lavage) or BAS (bronchoalveolar aspirate)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This multicentric, prospective study aims at:

evaluating the prevalence, etiology, characteristics, and 1one-year outcomes of immunocompromised patients hospitalized for Community-Acquired Pneumonia (CAP); conducting biochemical, microbiological and genetic analysis on collected samples.

DETAILED DESCRIPTION:
Primary endpoint:

Collection of in- hospitalisation mortality for all causes in immunocompromised patients with CAP enrolled.

Secondary endpoints:

Collection of data on admission and during hospitalisation to evaluate clinical response to empirical treatments (including antibiotic therapy) related to severity of disease and microbiological etiology.

Prevalence of cardiovascular events and all-cause mortality during hospitalization or after discharge.

Biochemical, microbiological and genetic analysis on collected samples.

ELIGIBILITY:
Inclusion Criteria:

Hospitalized patients with a confirmed diagnosis of Community-Acquired Pneumonia (CAP) characterized by at least one of the following risk factors for immunosuppression:

* AIDS,
* Aplastic anemia;
* Asplenia;
* Hematologic malignancy (e.g., lymphoma/acute or chronic myeloid leukemia/multiple myeloma);
* Chemotherapy within the last 3 months;
* Neutropenia defined as a white blood cell count less than 500/dL on a complete blood count;
* Use of biologics (including trastuzumab and therapy for autoimmune diseases (e.g., anti-TNF α), prescribed within the last 6 months before hospital admission;
* Solid organ transplant;
* Bone marrow transplant;
* Chronic oral steroid use (>10 mg/day prednisone or equivalent ≥3 months before accessing the ED, or cumulative dose > 600 mg prednisone);
* Use of corticosteroid therapy with a dose ≥ 20 mg prednisone or equivalent ≥14 days or cumulative dose > 600 mg prednisone;
* Active malignancy;
* Malignancy within one year of pneumonia (excluding patients with localized skin cancer or early-stage malignancy);
* Lung malignancy with neutropenia/chemotherapy;
* Other solid malignancy with neutropenia/chemotherapy;
* Other immunodeficiency (including congenital/genetic immunosuppression and immunosuppressive therapy secondary to hematologic malignancy or solid malignancy);
* Primary immunodeficiency.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Immunosuppressed patients with Community-Acquired Pneumonia will be enrolled during hospitalization in Italian Pneumology, Infectious Diseases and Emergency Departments selected on their specific experteeze and know-how. Upon discharge, patients will be followed up at 30 days, 3 months, 6 months and 12 months after discharge.
Sampling Method: Non-Probability Sample
Enrollment: 1298 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality for all causes in immunocompromised patients with CAP enrolled in the study. | During hospitalization corresponding to study enrollment (1 day to 2 weeks of hospitalization on average)
  Recording in-hospital mortality for all causes in immunocompromised patients with CAP enrolled in the study.

SECONDARY OUTCOMES:
Time to clinical stability | DAY 1 to 8
  Time to clinical stability calculated as the number of days from the date of admission to the date that the patient meets clinical stability criteria, up to 8 days. Clinical stability is defined as follows: improved clinical signs (improved cough and shortness of breath), lack of fever for at least 8 hours, improving leukocytosis (decreased at least 10% from the previous day), and tolerating oral intake.
Mortality for all causes in immunocompromised patients with CAP | 30 days, 3 months, 6 months and 12 months after hospital discharge.
  Mortality for all causes in immunocompromised patients with CAP enrolled in the study.
New hospitalizations in immunocompromised patients with CAP. | 30 days, 3 months, 6 months and 12 months after hospital discharge.
  Recording new hospitalizations in immunocompromised patients with CAP enrolled in the study.
Prevalence of cardiovascular events in immunocompromised patients with CAP. | 30 days, 3 months, 6 months and 12 months after hospital discharge.
  Prevalence of cardiovascular events in immunocompromised patients with CAP enrolled in the study.
Length of hospital stay (days) | Through hospital discharge, ranging from 1 day to 2 weeks
ICU admission % | During hospitalization corresponding to study enrollment (1 day to 2 weeks of hospitalization on average)
Need for mechanical ventilation % | During hospitalization (1 day to 2 weeks on average)
Lenght of mechanical ventilation (Hours) | During hospitalization (1 day to 2 weeks on average)
Rate of antibiotic therapy modification (%) | During hospitalization (1 day to 2 weeks on average)
Subsequent re-admission within 1 year | Within 365 days after hospital discharge
Characterization of Microbiological Etiology Using 16S rRNA Sequencing and Whole-Genome Sequencing | Through study completion, for up to 4 years
  Microbiological analysis will be performed on sputum, bronchoalveolar lavage (BAL), and bronchial aspirate (BAS) samples. The 16S rRNA sequencing will be conducted to evaluate the relative abundance of identified bacterial genera (percentage/total) and to calculate alpha diversity indices, including Shannon and Equitability indices. For samples where bacterial strains are isolated, whole-genome sequencing (WGS) will be performed to identify and study resistance, virulence, and pathogenicity genes. These findings will be correlated with clinical data to provide insights into microbiological etiology. Data will be summarized as relative abundances, diversity indices, and the presence/absence of key genomic features.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco B.A. Blasi, MD, Study Chair — Respiratory Unit and Cystic Fibrosis Center, Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico
Locations (1):
- Internal Medicine Department, Respiratory Unit and Cystic Fibrosis Center, Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico Milano Via Francesco Sforza 35 20122 Milan Italy, Milan, Milano, Italy

REFERENCES:
- [Background] Garcia-Vidal C, Fernandez-Sabe N, Carratala J, Diaz V, Verdaguer R, Dorca J, Manresa F, Gudiol F. Early mortality in patients with community-acquired pneumonia: causes and risk factors. Eur Respir J. 2008 Sep;32(3):733-9. doi: 10.1183/09031936.00128107. Epub 2008 May 28. PMID 18508820
- [Background] Metlay JP, Waterer GW, Long AC, Anzueto A, Brozek J, Crothers K, Cooley LA, Dean NC, Fine MJ, Flanders SA, Griffin MR, Metersky ML, Musher DM, Restrepo MI, Whitney CG. Diagnosis and Treatment of Adults with Community-acquired Pneumonia. An Official Clinical Practice Guideline of the American Thoracic Society and Infectious Diseases Society of America. Am J Respir Crit Care Med. 2019 Oct 1;200(7):e45-e67. doi: 10.1164/rccm.201908-1581ST. PMID 31573350
- [Background] Aliberti S, Cilloniz C, Chalmers JD, Zanaboni AM, Cosentini R, Tarsia P, Pesci A, Blasi F, Torres A. Multidrug-resistant pathogens in hospitalised patients coming from the community with pneumonia: a European perspective. Thorax. 2013 Nov;68(11):997-9. doi: 10.1136/thoraxjnl-2013-203384. Epub 2013 Jun 17. PMID 23774884
- [Background] Evans SE, Ost DE. Pneumonia in the neutropenic cancer patient. Curr Opin Pulm Med. 2015 May;21(3):260-71. doi: 10.1097/MCP.0000000000000156. PMID 25784246
- [Background] Feldman C. Pneumonia associated with HIV infection. Curr Opin Infect Dis. 2005 Apr;18(2):165-70. doi: 10.1097/01.qco.0000160907.79437.5a. PMID 15735422
- [Background] Di Pasquale MF, Sotgiu G, Gramegna A, Radovanovic D, Terraneo S, Reyes LF, Rupp J, Gonzalez Del Castillo J, Blasi F, Aliberti S, Restrepo MI; GLIMP Investigators. Prevalence and Etiology of Community-acquired Pneumonia in Immunocompromised Patients. Clin Infect Dis. 2019 Apr 24;68(9):1482-1493. doi: 10.1093/cid/ciy723. PMID 31222287
- [Background] Carugati M, Aliberti S, Sotgiu G, Blasi F, Gori A, Menendez R, Encheva M, Gallego M, Leuschner P, Ruiz-Buitrago S, Battaglia S, Fantini R, Pascual-Guardia S, Marin-Corral J, Restrepo MI; GLIMP Collaborators. Bacterial etiology of community-acquired pneumonia in immunocompetent hospitalized patients and appropriateness of empirical treatment recommendations: an international point-prevalence study. Eur J Clin Microbiol Infect Dis. 2020 Aug;39(8):1513-1525. doi: 10.1007/s10096-020-03870-3. Epub 2020 Apr 3. PMID 32242314
- [Background] Ramirez JA, Musher DM, Evans SE, Dela Cruz C, Crothers KA, Hage CA, Aliberti S, Anzueto A, Arancibia F, Arnold F, Azoulay E, Blasi F, Bordon J, Burdette S, Cao B, Cavallazzi R, Chalmers J, Charles P, Chastre J, Claessens YE, Dean N, Duval X, Fartoukh M, Feldman C, File T, Froes F, Furmanek S, Gnoni M, Lopardo G, Luna C, Maruyama T, Menendez R, Metersky M, Mildvan D, Mortensen E, Niederman MS, Pletz M, Rello J, Restrepo MI, Shindo Y, Torres A, Waterer G, Webb B, Welte T, Witzenrath M, Wunderink R. Treatment of Community-Acquired Pneumonia in Immunocompromised Adults: A Consensus Statement Regarding Initial Strategies. Chest. 2020 Nov;158(5):1896-1911. doi: 10.1016/j.chest.2020.05.598. Epub 2020 Jun 16. PMID 32561442